CLINICAL TRIAL: NCT02502578
Title: Phase I/IIa Study of CNT-01 in Patients With Idiopathic Triglyceride Deposit
Brief Title: Safety Study of CNT-01 in Patients With Idiopathic TGCV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Osaka University (Other)
Responsible Party: Principal Investigator, Ken-ichi Hirano, Assistant Professor, Osaka University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNT-01-001
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Idiopathic Triglyceride Deposit Cardiomyovasculopathy
Keywords: Triglyceride Deposit Cardiomyovasculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CNT-01 (Experimental): Patients will receive CNT-01 500 mg orally three times daily for 14 days. On Day 15, patients will take CNT-01 500 mg only once after blood drawing.
  Interventions: Drug: CNT-01 500 mg capsule

INTERVENTIONS:
Drug: CNT-01 500 mg capsule — After being informed about the study and potential risks, all patients giving written informed consent undergo screening tests to determine eligibility for study enrollment. On Day 1, patients who meet the eligibility criteria will start taking CNT-01 500mg orally three times daily for 14 days. On Day 15, patients will take CNT-01 500 mg only once after blood drawing.

SUMMARY:
The purpose of this study is to assess the safety and to examine the index of the efficacy after repeated dosing of CNT-01 in patients with idiopathic triglyceride deposit cardiomyovasculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Have a definite diagnosis of idiopathic triglyceride deposit cardiomyovasculopathy
* After receiving a sufficient explanation upon participation in this study, on a full understanding, patients who obtained the written informed consent from each patient
* More than 20 years old at the time of informed consent
* Is able to oral intake
* Must be willing to comply with protocol-required examination such as BMIPP myocardial scintigraphy

Exclusion Criteria:

* Have diabetic ketoacidosis
* Have a malignancy that is being treated by anticancer drug or anticipated survival is less than three years
* Female with pregnant or lactating
* Is not able to agree to using intrauterine device, oral contraceptive, condom or having sexual intercourse from the start of taking investigational product to 30 days after the end of the study
* Have a New York Heart Association functional classification IV
* Have a known history of drug dependence
* Is allergic to any component of the investigational product
* Is allergic to BMIPP or iodine
* Have a known history of clinically significant drug allergy
* Have a severe liver dysfunction (Child classification B and C)
* Participated in other clinical study within the past 3 months and received an investigational agent including placebo
* Being treated with diet containing medium chain fatty acid
* Is considered unfit for the study by the Investigator's medical decision

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of adverse event | Baseline to Day 29
Change in 12-lead ECG recordings from Baseline | Baseline to Day 29
Change in Blood Pressure from Baseline | Baseline to Day 29
Change in clinical laboratory testings as measured by serum chemistry, hematology and urinalysis from Baseline (composite) | Baseline to Day 29
Change in Body temperature from Baseline | Baseline to Day 29
Change in Pulse rate from Baseline | Baseline to Day 29

SECONDARY OUTCOMES:
Change in uptake and washout rate in BMIPP myocardial scintigraphy | Baseline to Day 15
Change in blood concentration of fatty acid fraction from Baseline (Octanoic acid, Capric acid, Myristic acid, Palmitic acid and Stearic acid) | Baseline to Day 16
Change in lipase activity in peripheral polynuclear leucocyte from Baseline | Baseline to Day 29
Change in blood lipoprotein fraction from Baseline | Baseline to Day 29
Change in vacuolation rate in polynuclear leucocyte from Baseline | Baseline to Day 29
Change in frequency in use of nitroglycerin from Baseline | Baseline to Day 29
Change in New York Heart Association (NYHA) functional classification from Baseline | Baseline to Day 29
Change in reactive hyperemic index from Baseline | Baseline to Day 29
Change in score of SF-36 from Baseline | Baseline to Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Ken-ichi Hirano, M.D., Ph.D., Study Chair — Department of Cardiovascular Medicine, Osaka University Graduate School of Medicine
Locations (1):
- Cardiovascular Medicine, Osaka University Hospital, Suita, Osaka, Japan